CLINICAL TRIAL: NCT07217483
Title: The Feasibility of Prolacta CR for Treatment of Neonatal Hypoglycemia
Brief Title: The Feasibility of Cream for Treatment of Neonatal Hypoglycemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 023-279
Record Dates: First submitted 2025-10-12; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Neonatal Hypoglycemia

STUDY DESIGN:
Intervention Model Description: In this study the newborns with low blood glucose, but have no symptoms, will be managed by giving 3 ml/kg of Prolact CR (cream) instead of 0.5 ml/kg of 40% oral dextrose gel. Blood glucose will be monitored one hour after the cream is given. If needed, according to the protocol baby will receive up to three doses of cream. If baby has symptoms with low blood glucose, will receive intravenous dextrose.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Prolact CR (Other): One arm receiving Prolact CR for hypoglycemia
  Interventions: Dietary Supplement: Prolact CR for hypoglycemia

INTERVENTIONS:
Dietary Supplement: Prolact CR for hypoglycemia — Utilizing Prolact CR instead of dextrose gel for management of newborn hypoglycemia

SUMMARY:
Prolact CR (cream) is a fat supplement that is derived from pasteurized human donor milk. It has been utilized in babies who are born premature in the neonatal intensive care unit (NICU) setting to improve growth while avoiding cow milk exposure. There is no literature on the use of cream as a treatment for low blood glucose levels in newborns who are at risk. It is known that fat in human colostrum plays a vital role in providing energy, substrate, and stimulates gluconeogenesis. Gluconeogenesis is the process that helps in the sustainment of blood glucose. Dextrose gel that is used to treat low blood glucose levels helps in raising the blood glucose, but does not help in sustainment.

The objective of this pilot study is to evaluate the utility, feasibility, and acceptability of administering cream for the treatment of newborn low blood glucose levels in a couplet care unit. Investigators hypothesized that 3 ml/kg of cream (0.2 g/kg of carbohydrate and 0.75 g/kg of fat), if given in the place of 0.5 ml/kg (0.2 g/kg of carbohydrate) would increase and stabilize the blood glucose levels. Investigators also speculated that newborns would tolerate the cream with no adverse effects, and caregivers (nurses and parents) would find its use feasible and acceptable.

Parents of newborns with risk factors for hypoglycemia [born to mothers with diabetes, small for gestational age, large for gestational age, or late prematurity (35 to 37 weeks' gestation at birth) who intended to breastfeed exclusively will be approached to consent for the study either before or after delivery of the infant. Newborns with major congenital anomalies or those admitted immediately to the NICU after birth will be excluded.

The main questions hoping to answer

1. What percentage of newborns receiving cream for treatment of hypoglycemia will need NICU admission for IV dextrose?
2. How many median doses of cream are needed?
3. What percentage of infants will be discharge exclusively feeding human milk from couplet care unit?
4. What percentage of the surveys will show parent/nursing satisfaction with the product?

ELIGIBILITY:
Inclusion Criteria:

* Newborns at risk for hypoglycemia (born to mothers with diabetes, small for gestational age, large for gestational age, late preterm born 35 to 37 weeks gestational age)

Exclusion Criteria:

* Newborns with major congenital anomalies
* Newborns directly admitted to the NICU form delivery room

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
NICU admission | Birth to hospital discharge at 2 to 5 days of life
  Admission to neonatal intensive care unit for intravenous dextrose for treatment of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Arpitha Chiruvolu, MD, Study Chair — Baylor Scott & White Medical Center - McKinney
Locations (1):
- Baylor Scott & White Medical Center - McKinney, McKinney, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT07217483/ICF_000.pdf